CLINICAL TRIAL: NCT02679872
Title: Important Non-technical Skills When Performing Video-assisted Thoracoscopic Surgery: Perceptions of the Operating Team
Brief Title: Video-assisted Thoracoscopic Surgery Teams' Perception of Non-technical Skills
Status: Completed | Type: Observational
Sponsor: Copenhagen Academy for Medical Education and Simulation (Other)
Responsible Party: Principal Investigator, Kirsten Gjeraa, PhD student, medical doctor., Copenhagen Academy for Medical Education and Simulation
Other Study IDs: R100-A7166
Record Dates: First submitted 2016-02-04; First posted 2016-02-10 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Lung Cancer
Keywords: Non-technical skills; Patient safety; Video-assisted thoracoscopic surgery; Operating theatre team; Operating room
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- VATS team 1: Video-assisted thoracoscopic surgery team, from institution/hospital 1.
- VATS team 2: Video-assisted thoracoscopic surgery team, from institution/hospital 2.
- VATS team 3: Video-assisted thoracoscopic surgery team, from institution/hospital 3.
- VATS team 4: Video-assisted thoracoscopic surgery team, from institution/hospital 4.

SUMMARY:
Good non-technical skills (NTS) have been shown to prevent adverse events and errors. Improvements of NTS can be achieved by simulation based-team training.The NTS of the operating theatre team performing video-assisted thoracoscopic surgery (VATS) is speculated to differ fra open thoracic surgery, as is the case with technical skills; however, these have not been investigated. The aim of this study is to explore which NTS the members of the VATS team perceive to be most important to patient care and safety. Exploration will be done through a deductive, qualitative analysis of semi-structured group and individual interviews with VATS team members. A theoretical perspective of Hollnagels Safety-II will be taken using the taxonomy of Oxford Non-Technical Skills (NOTECHS) system with the aim of informing patient safety.

DETAILED DESCRIPTION:
BACKGROUND:

Non-technical skills (NTS) can be defined as 'the cognitive, social and personal resource skills that complement technical skills, and contribute to safe and efficient task performance'. Human errors, such as communication breakdowns, lack of speaking up and of good leadership, are known to contribute considerably to adverse events. Adverse events are common in the operating theatre affecting patient safety. Adaptive behaviours have been shown important as a response to the dynamic, complex world of the operating theatre to prevent potential problems and adverse events.

As with technical skills, NTS can be taught by team training. Team training have been shown to improve attitudes as well as NTS, and reduced technical errors. Large studies have additionally shown that team training can reduce adverse events and improve patient outcome. A training intervention targeted at operating theatre teams will need to start with an assessment uncovering the learning needs of the team members.

In general minimally invasive surgery (MIS) is shown to be more complex, involve more personnel and take longer time than open surgery. The technical skills are different, among other things due to complex equipment and two-dimensional vision of a three-dimensional operating space. In our systematic review (submitted), only few studies investigated the NTS in MIS teams. The communication in MIS compared to open surgery were found to be different, relating more to equipment and patient related topics. Working in fixed teams improved teamwork climate in MIS teams.

Correspondingly, the NTS of the video-assisted thoracoscopic surgery (VATS) operating team is speculated to differ from the NTS needed in open surgery as is the case with the technical skills. However, no studies investigated the NTS of VATS teams.

The aim of this study is to explore, which NTS the members of the VATS team perceive to be most important to high quality patient care and patient safety.

METHODS:

Frameworks/theory:

The theoretical conceptual framework for the study is the safety theory by Erik Hollnagel, named Safety-I and Safety-II, arguing for a new view on safety: Safety-II. In Safety-I, the ontology is that things either function or malfunction, that could be a piece of equipment or healthcare professionals following procedures or guidelines. Consequently, the aetiology of the outcomes can be explained by a cause-effect relationship, where the malfunction of things linearly cause an unwanted effect. The resulting phenomenology then refers to outcomes as adverse events / incidents/ accidents. Oppositely, in Safety-II, the ontology is that in socio-technical systems, such as the healthcare system, performance adjustments is needed to adjust work, that is the task and the tools, to the actual situation of the complex world. Hence, as the technology only can vary to a limited extent, human performance needs to vary. The aetiological explanation in Safety-II is therefore, that performance variability resonate through both proactive and reactive adjustments into observed outcomes, named emergent outcomes. The resulting phenomenology sees the performance variability as both the basis of adverse events and of acceptable outcomes; that is everyday activities. These performance adjustments can be categorised into three types of adjustments: Maintaining/creating, compensating and avoiding, thereby characterising the performance variability for a specific activity. In all, the starting point is turned around. In Safety-II, the focus is on why and how things go right with the aim of understanding everyday activities, termed 'Work-as-Done', in contrast to the less interesting written procedure guidelines etc., termed 'Work-as-Imagined'.

Within non-technical skills research and education in healthcare, and especially within the specialities working in the operating theatre, a taxonomy widely used is the framework of behavioural markers adapted from the aviation industry, termed the Oxford Non-Technical Skills (NOTECHS) system. This framework is structured around four categories, divided into several elements each represented by examples of good or poor behavioural markers. This system has been developed and evaluated for operating teams and assesses both the team and each subteam's NTS. In this study, the taxonomy of the NOTECHS system in the perspective of the conceptual theory of Safety-II will be used as framework for the data analysis as described in detail below. In all, the behavioural markers representing good behaviours will therefore be the focus of this study to explore how things go right as this is much often the case than not. Interviewing the actual VATS team members themselves will explore their own perception of the NTS used in their everyday activities including the needed adaptions to situational requirements, found by others. This will represent 'Work-as-Done' rather than 'Work-as-Imagined' with the aim of informing the Safety-II perspective on patient safety.

Design:

The study will use the theories described above in an explorative semi-structured interview study. The data collection and thereby sample size will be an iterative process until no new data is revealed, hence saturation is met. This will include interviews of both multi-professional teams and individuals depending on the data revealed during the interviewing-analysing process. Interviews will be conducted by KG and ASM using a semi-structured interview guide. The interview guide will be adjusted during the iterative process of interviews and analysis. All interviews will be audio-recorded and transcribed verbatim. The study will be reported in accordance with the Standards for Reporting Qualitative Research (SRQR). Quality and rigour will be aimed for as suggested for qualitative research.

Ethics:

The Regional Scientific Ethics Committee of the Capital Region will be applied; however, we expect a letter of exemption due to Danish laws on educational studies not involving patients. Participants will receive oral and written information and will have to give informed consent with the continuous option of retracting their consent and participation. Personal data will be stored according to Danish Data Protection Law, and will be presented anonymously. The study protocol will be registered at www.clinicaltrials.gov.

Participants, setting and time:

Participants will be purposefully sampled as subject matter experts in terms of VATS operating teams in conjunction with individuals. The teams will consist of one or two surgeon(s) with VATS experience, one younger assisting surgeon, one anaesthesiologist, one nurse anaesthetist, and one to two scrub nurses with experience as both assisting and circulating nurse. The individuals will be relevant healthcare professionals of any of the above. Participants will come from the four university hospitals performing VATS in Denmark in collaboration with head of departments. Each person will only be included in one team interview and/or one individual interview. The interviews are planned to be conducted in February and March 2016.

The interview guide:

The interview guide will be semi-structured with a scripted introduction before each interview setting the scene and the topic of the interview. The interview will try to explore all four NOTECHS categories, namely leadership & management, teamwork & co-operation, problem-solving & decision-making, and situation awareness in a Safety-II perspective, focusing on the performance variability of the team members needed in their daily work to adapt to situational requirements. Emphasis will be laid on allowing all team members to give their perspective in order to explore views of the entire team. The interviews will be semi-structured so probe questions will be used when necessary to obtain additional information.

Prior to conducting the interviews, two authors (KG, ASM) will spend a number of hours observing VATS procedures in order to become familiar with the procedures and with any critical phases of the operations. This, along with input from experienced VATS surgeons (RHP, HJH) and an experienced anaesthesiologist (DO), will inform the interview guide. The interview guide will be internally reviewed by the authors consisting of surgeons, a scrub nurse and an anaesthesiologist that are experienced qualitative and NTS researchers. It will be pilot tested on healthcare professionals without specific NTS knowledge to avoid misunderstanding and misinterpretation; however, these data will not be included in the study.

Data collection and analysis:

The interviews will be conducted face-to-face in undisturbed rooms in relation to the operating theatre in or just after normal working hours depending on working schedule. The participants demographic data will be collected consisting of profession, age, gender, years of clinical experience, years and type of experience with laparoscopic or VATS procedures and previous experience with NTS training.

A deductive data analysis strategy will be applied in this study. With the taxonomy of the NOTECHS framework we will use directed content analysis to analyse the interviews. Directed content analysis can be applied when 'prior research exists about a phenomenon that is incomplete/would benefit from further description'. As we approach the topic from a Safety-II perspective, focus will be on which behaviours the VATS team members perceive as important in insuring that things go right thereby insuring high quality patient care and patient safety. Explicitly we will focus on performance variability in their everyday work, categorising them as either maintaining/creating, compensating or avoiding.

The strategy is to use the categories of NOTECHS as well as categories of performance variability, when reading the transcribed interviews. The text will then be coded into these categories for condensation, adding new ones when extra text of interest is uncovered in order to avoid missing important new information that could inform the theory on NTS in VATS teams. The text coded will be marked to adhere to one of the categories, introducing new categories if needed. The texts will then be paraphrased to condense the interview quotations into observable behavioural examples.

The analyses will be conducted by KG and ASM. The first interviews will be coded by both KG and ASM; the coding will be discussed between these two and LS/DO. When agreement is satisfactorily, the two authors will split up and code the remaining interviews independently. The results of the coding will be discussed with LS/DO and later the full group of authors. The analysis will be conducted using NVivo (version 10).

Acknowledgements:

The authors will like to thanks the participating cardiothoracic departments in Denmark.

PROJECT ORGANISATION:

This study will be conducted at Copenhagen Academy for Medical Education and Simulation (CAMES), at Rigshospitalet, Capital Region of Denmark and Copenhagen University.

Members of the research group:

Project leader, MD, PhD student Kirsten Gjeraa (KG) Interviewer and analyser, CRN Anna Sofie Mundt (ASM) Co-supervisor, MD, PhD Lene Spanager (LS) Co-supervisor, MD Henrik Jessen Hansen (HJH) Co-supervisor, MD René Horsleben Petersen (RHP) Co-supervisor, MD, PhD, associate professor Lars Konge (LK) Supervisor, MD, DMSc, MHPE, professor Doris Østergaard (DO)

Publication:

The results will be published in an international journal.

Author list:

Kirsten Gjeraa, Anna Sofie Mundt, Lene Spanager, Lars Konge, René Horsleben Petersen, Henrik Jessen Hansen, Doris Østergaard.

ELIGIBILITY:
Inclusion Criteria:

* Medical doctors and medical nurses with experience in VATS by purposeful sampling.

Exclusion Criteria:

* Medical doctors and medical nurses with experience in VATS, who are included in the project group of the present study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Medical doctors, medical nurses with experience in VATS
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2016-02; Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Transcribed interviews | 3 months
  Group interviews, and individual interviews if nessesary, with the VATS team members.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] REFERENCE LIST: upon request.
- Available data/document: Study Protocol — http://www.regionh.dk/CAMES — Possible to request full protocol, inclusive full reference list, in pdf from first investigator Kirsten Gjeraa, MD, email: kirsten.gjeraa@regionh.dk